CLINICAL TRIAL: NCT02594631
Title: Shock Wave Lithotripsy Versus Visual Cystolitholapaxy in The Management of Patients Presenting With Calcular Acute Urinary Retention: A Randomized Controlled Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Ali, Resident in Urology, Urology and Nephrology Center, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MALI1112015
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Calculi
Keywords: Urethral stones; Acute Cacular urinary retention; Extracorporeal Shock Wave Lithotripsy (ESWL); Visual lithotripsy; bladder stone
MeSH Terms: conditions — Urinary Calculi; Urinary Bladder Calculi | interventions — Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESWL Group (Active Comparator): Patients in this arm will receive ESWL as treatment for acute calcular urinary retention
  Interventions: Procedure: ESWL
- Endoscopy group (Active Comparator): Patients in this arm will receive endoscopic treatment for acute calcular urinary retention
  Interventions: Procedure: Endoscopic treatment

INTERVENTIONS:
Procedure: ESWL — Patients in this arm will receive ESWL for treatment of acute calcular urinary retention
  Other Names: Extracorporeal shock wave lithotripsy
  Arms: ESWL Group
Procedure: Endoscopic treatment — Patients in this arm will receive endoscopic treatment of acute calcular urinary retention
  Other Names: Visual litholapaxy
  Arms: Endoscopy group

SUMMARY:
The aim of the study is to compare the safety and efficacy of ESWL and visual cystolitholapaxy in management of calcular acute urine retention.

DETAILED DESCRIPTION:
Patients who present with acute urinary retention due to stone in the urethra or urinary bladder will be randomly assigned to receive treatment either by extracorporeal shock wave lithotripsy or by endoscopic visual cystolitholapaxy where patients and stone characteristics will be recorded and the outcome including the intraoperative and postoperative complications and the stone free rate will be also evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients presenting with acute urinary retention due to urethral or urinary bladder stones.
2. with a stone size not more than 2 centimeters in greatest diameter.
3. No more than 2 stones.

Exclusion Criteria:

1. Bladder cancer.
2. Bladder replacement of any type.
3. Infravesical obstruction, due to marked benign prostatic hyperplasia, prostate cancer, stricture urethra or external urethral meatal stenosis.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 1 week
  evaluation of stone free rate after the assigned intevention

SECONDARY OUTCOMES:
Adverse events after the assigned intervention | 1 month
  evaluation of adverse events after the assigned intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Shokeir, Prof, Study Chair — Urology and Nephrology Cenetr
Locations (1):
- Urology an Nephrology Center, Al Mansurah, DK, Egypt